CLINICAL TRIAL: NCT01961960
Title: Phase 3 Study of ASP7374 -Open-label Study of Intramuscular ASP7374 in Adults ≥61 Years of Age-
Brief Title: A Study to Evaluate Intramuscular ASP7374
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMN Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 7374-CL-0105
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Influenza; Vaccine
Keywords: ASP7374; Prevention of seasonal influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP7374 group (Experimental)
  Interventions: Biological: ASP7374

INTERVENTIONS:
Biological: ASP7374 — intramuscular

SUMMARY:
The purpose of this study is to evaluate safety and immunogenicity of intramuscular ASP7374 in adults ≥61 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or medically stable, as judged on the basis of history and concurrent diseases.
* Subject understands procedure of the protocol and is willing to comply with the protocol.
* Written informed consent has been obtained.

Exclusion Criteria:

* Scheduled to receive another vaccine during the study.
* Received influenza HA vaccine within 180 days prior to screening.
* Received or scheduled to receive a live vaccine within 28 days prior to vaccination with the study vaccine, and received or scheduled to receive an inactivated vaccine or a toxoid within 7 days prior to vaccination with the study vaccine.
* Diagnosis of immune deficit in the past, has a family member (within the third degree of kinship) with a diagnosis of congenital immunodeficiency syndrome.
* Received one of the following medications or treatment prior to vaccination with the study vaccine: Interferon formulation, Drugs which affect the immune system, corticosteroids, G-CSF, M-CSF, Human immunoglobulin products, Blood products, Blood transfusion
* History of anaphylactic shock or an allergic reaction such as generalized eruption due to food or drug (including vaccines) allergies, fever ≥39.0°C within 2 days after the previous vaccination (influenza vaccine and others)
* History of seizures, except for febrile seizures in childhood

Min Age: 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
hemagglutination inhibition (HI) antibody titer | Day 1 and Day 29
  evaluated for A/H1N1, A/H3N2, and B

SECONDARY OUTCOMES:
neutralizing antibody titer | Day 1 and Day 29
  evaluated for A/H1N1, A/H3N2, and B
Local and systemic reactions associated with the vaccination | Day 1 through Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Principal Investigator — Astellas Pharma Inc
Locations (1):
- Kanto, Japan